CLINICAL TRIAL: NCT00606996
Title: Group IPT for Women Prisoners With Comorbid Substance Use and Depression
Brief Title: Group Therapy for Women Prisoners With Comorbid Substance Use and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Johnson, Associate Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23DA021159-01 (NIH); NCT01831349 (obsolete NCT alias)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Substance Abuse; Substance Dependence; Depressive Disorder
Keywords: Drug Abuse; Drug Dependence; Alcohol Abuse; Alcohol Dependence; Major Depressive Disorder; Dysthymic Disorder; Prisoners; Women
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder; Alcoholism; Depressive Disorder, Major; Dysthymic Disorder

ARMS (2):
- IPT-G (Experimental): Group Interpersonal Psychotherapy
  Interventions: Behavioral: Group interpersonal psychotherapy (IPT-G)
- PSYCHOED (Active Comparator): Psychoeducation
  Interventions: Behavioral: Psychoeducation on co-occurring disorders (PSYCHOED)

INTERVENTIONS:
Behavioral: Group interpersonal psychotherapy (IPT-G)
  Arms: IPT-G
Behavioral: Psychoeducation on co-occurring disorders (PSYCHOED)
  Arms: PSYCHOED

SUMMARY:
The purpose of the study is to determine whether interpersonal psychotherapy is effective for treating co-occurring depression and substance use among women prisoners.

DETAILED DESCRIPTION:
Incarcerated women are a vulnerable and rapidly expanding population with high lifetime rates of both substance use disorder (SUD; abuse or dependence on alcohol, illegal drugs, or prescription drugs; 70%) and depressive disorder (DD; major depressive disorder and dysthymic disorder; 20-27%). DDs tend to worsen the course of SUDs for incarcerated women by increasing their risk for suicide attempts, contributing to the persistence of substance abuse, and reducing the likelihood of a successful transition to an independent, sober life in the community. Recent evidence indicates that DDs are common in persons with SUDs, often do not remit with SUD treatment, and should be treated. Despite growing recognition that co-occurring disorders, such as DDs, among substance abusing incarcerated women present an important public health concern, integrated treatments for SUD-DD have not been well-developed for or systematically tested in this population. Group Interpersonal Psychotherapy (IPT-G) has been shown to be efficacious in treating DD in other populations and may be especially pertinent to the needs of incarcerated women with SUD-DD because interpersonal difficulties not only affect severity of depression, but are also strong predictors of drinking to cope, SUD relapse, and prison recidivism in women.

This study tests the hypotheses that as adjuncts to prison SUD treatment, IPT-G, relative to psychoeducation on co-occurring disorders, will produce at least moderate effect sizes for:

* Reduction in the risk and severity of substance use relapse after release from prison
* Recovery from depressive disorder and reduction in depressive symptoms
* Improvement in social support and interpersonal functioning
* Reduction in the severity of legal problems during the 3 month follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Participants are recruited from prison substance use treatment programs.
* Current primary (non-substance-induced, as defined by the SCID) depressive disorder (major depressive or dysthymic disorder) after at least 4 weeks of prison SUD treatment and abstinence.
* A minimum Hamilton Depression score of 18 or higher, indicating moderate to severe depression.
* Depressive disorder at any time while not incarcerated.
* Substance use disorder one month prior to incarceration.
* Between 10 and 18 weeks away from release from prison.

Exclusion Criteria:

* Lifetime criteria for bipolar disorder
* Lifetime criteria for a psychotic disorder
* Actively suicidal

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Substance-free days after release from prison, measured by the Timeline Followback method | 3 months post-release
Severity of substance use after release from prison, measured by the Addiction Severity Index | 3 months post-release
Verification of substance-free status using breath alcohol tests and urine drug screens | 3 months post-release
Depression symptom severity measured by the Modified Hamilton Rating Scale for Depression | Pre-release
Depression symptom severity measured by the Beck Depression Inventory | Pre-release

SECONDARY OUTCOMES:
Severity of legal problems after release, measured by the Legal Composite of the Addiction Severity Index | 3 months post-release
Interpersonal problems, measured by the Inventory of Interpersonal Problems | 3 months post-release
Peer support and social support, measured by the Criminal Justice client Evaluation of Self and Treatment | 3 months post-release
Perceived social support measured by the Multidimensional Scale of Perceived Social Support | 3 months post-release
Social support for recovery, measured by the Important People and Activities scale | 3 months post-release
Social functioning, measured by the Social Adjustment Scale | 3 months post-release

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Johnson, Ph.D., Principal Investigator — Department of Psychiatry and Human Behavior, Brown University
Locations (1):
- Adult Correctional Institution, Cranston, Rhode Island, United States